CLINICAL TRIAL: NCT00887952
Title: Alternative Treatment of Deep Caries Lesions Based on Biological Evidences
Brief Title: Partial Removal of Caries Dentines
Acronym: PRCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Ivoclar Vivadent AG (Industry)
Responsible Party: Marisa Maltz, Odontology Faculty - Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FO UFRGS; FAPERGS 04/1531.8; CNPQ 403420/04
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-04

CONDITIONS: Dental Caries
Keywords: Deep caries lesion; dentine caries removal; dental restoration; stepwise excavation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Partial removal of carious dentine. Carious dentine partial removal plus restoration in one session. The group is divided according to the filling material: amalgam or resin.
  Interventions: Procedure: Partial removal of carious dentine
- 2 (Active Comparator): Stepwise excavation: Carious dentine removal performed in 2 steps: partial removal of carious dentine, indirect pulp capping (calcium hydroxide cement); temporary filling with IRM; cavity re-opening after 60 days, removal of the remaining soft carious tissue and filling (amalgam or resin).
  Interventions: Procedure: Stepwise excavation

INTERVENTIONS:
Procedure: Partial removal of carious dentine — All procedures will be carrying out under local anesthesia and rubber dam. The treatment will be performed as follow: access to the lesion using rotator instruments (if necessary); fully removal of carious tissue from the cavity walls according to hardness criteria by rotator instruments and/or hand excavator; removal of the necrotic carious tissue (soft and disorganized carious tissue) from the cavity floor by hand excavator (to avoid pulp exposure); cleaning with distilled water and drying with sterile filter paper; group randomization. If the tooth is assigned to test group: cavity floor covered with calcium hydroxide cement; restoration using amalgam or steel crown following their usual clinical procedures based on the instructions of the manufacturer
  Arms: 1
Procedure: Stepwise excavation — The treatment will be performed as follow: access to the lesion using rotator instruments (if necessary); fully removal of carious tissue from the cavity walls according to hardness criteria by rotator instruments and/or hand excavator; removal of the necrotic carious tissue (soft and disorganized carious tissue) from the cavity floor by hand excavator (to avoid pulp exposure); cleaning with distilled water and drying with sterile filter paper; group randomization. If the tooth is assigned to SE: indirect pulp capping with calcium hydroxide cement; temporary filling with IRM; cavity re-opening after 60 days, removal of the remaining soft carious tissue and filling following the same procedures described to test group.
  Arms: 2

SUMMARY:
The aim of this multicenter randomized controlled clinical trial is to evaluate the effectiveness of an alternative treatment for deep caries lesions in Public Health Services. The alternative treatment consists of partial removal of carious dentine followed by restoration. The subjects were assigned to test or control groups: test - carious dentine partial removal and restoration in one session, and control - stepwise excavation. The stepwise excavation consists of partial removal of carious tissue from the cavity floor, indirect pulp capping with calcium hydroxide cement; temporary filling; cavity re-opening after 60 days, removal of the remaining soft carious tissue and filling. Each group was divided according to the filling material: amalgam or resin. The radiological exams are being performed before and after the treatment and then annually. Clinical evaluation of the restorations is performed right after the treatment and then annually (modified USPHS System). All evaluations are performed by calibrated and trained dentists.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ nine years old;
* permanent molars with primary deep caries lesion reaching dentine inner half (radiographic exam);
* pulpal sensibility positive (cold test);
* absence of spontaneous pain;
* absence of periapical alterations (radiographic exam);
* negative percussion test.

Exclusion Criteria:

* subjects with general diseases affecting their caries experience;
* caries lesion evolving an entire cusp;
* caries lesion with cervical margin in dentine.

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 329 (Actual)
Dates: Start 2005-08; Primary Completion 2008-11 (Actual); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Pulp sensitivity | Once a year during at least five years

SECONDARY OUTCOMES:
Remineralization of the residual caries (measure through digital substraction of radiographic exams) | Once a year during at least five years
Cost-effectiveness analysis | During five years of follow-up
Clinical evaluation of amalgam and resin restorations (USPHS criteria) | Once a year during at least five years

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Maltz, PhD, Principal Investigator — Odontology Faculty - Federal University of Rio Grande do Sul; Heliana Mestrinho, PhD, Study Chair — Odontology Faculty - Federal University of Brasília; Lilian M De Paula, PhD, Study Chair — Odontology Faculty - Federal University of Brasília; Juliana J Jardim, MSc, Study Chair — Odontology Faculty - Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Odontology Faculty - Federal University of Brasília, Brasília, Federal District
  - Odontology Faculty - Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Maltz M, Oliveira EF, Fontanella V, Carminatti G. Deep caries lesions after incomplete dentine caries removal: 40-month follow-up study. Caries Res. 2007;41(6):493-6. doi: 10.1159/000109349. Epub 2007 Oct 5. PMID 17921671
- [Background] Oliveira EF, Carminatti G, Fontanella V, Maltz M. The monitoring of deep caries lesions after incomplete dentine caries removal: results after 14-18 months. Clin Oral Investig. 2006 Jun;10(2):134-9. doi: 10.1007/s00784-006-0033-8. Epub 2006 Mar 21. PMID 16550396
- [Background] Maltz M, de Oliveira EF, Fontanella V, Bianchi R. A clinical, microbiologic, and radiographic study of deep caries lesions after incomplete caries removal. Quintessence Int. 2002 Feb;33(2):151-9. PMID 11890029
- [Background] Mertz-Fairhurst EJ, Curtis JW Jr, Ergle JW, Rueggeberg FA, Adair SM. Ultraconservative and cariostatic sealed restorations: results at year 10. J Am Dent Assoc. 1998 Jan;129(1):55-66. doi: 10.14219/jada.archive.1998.0022. PMID 9448347
- [Background] Bjorndal L. Indirect pulp therapy and stepwise excavation. J Endod. 2008 Jul;34(7 Suppl):S29-33. doi: 10.1016/j.joen.2008.02.035. PMID 18565369
- [Background] Bjorndal L, Larsen T. Changes in the cultivable flora in deep carious lesions following a stepwise excavation procedure. Caries Res. 2000 Nov-Dec;34(6):502-8. doi: 10.1159/000016631. PMID 11093026
- [Background] Bjorndal L, Thylstrup A. A practice-based study on stepwise excavation of deep carious lesions in permanent teeth: a 1-year follow-up study. Community Dent Oral Epidemiol. 1998 Apr;26(2):122-8. doi: 10.1111/j.1600-0528.1998.tb01938.x. PMID 9645406
- [Background] Ricketts DN, Kidd EA, Innes N, Clarkson J. Complete or ultraconservative removal of decayed tissue in unfilled teeth. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD003808. doi: 10.1002/14651858.CD003808.pub2. PMID 16856019
- [Derived] Jardim JJ, Mestrinho HD, Koppe B, de Paula LM, Alves LS, Yamaguti PM, Almeida JCF, Maltz M. Restorations after selective caries removal: 5-Year randomized trial. J Dent. 2020 Aug;99:103416. doi: 10.1016/j.jdent.2020.103416. Epub 2020 Jun 22. PMID 32585263
- [Derived] Maltz M, Garcia R, Jardim JJ, de Paula LM, Yamaguti PM, Moura MS, Garcia F, Nascimento C, Oliveira A, Mestrinho HD. Randomized trial of partial vs. stepwise caries removal: 3-year follow-up. J Dent Res. 2012 Nov;91(11):1026-31. doi: 10.1177/0022034512460403. Epub 2012 Sep 14. PMID 22983407